CLINICAL TRIAL: NCT04166929
Title: Haploidentical Stem Cell Transplantation With or Without NK Cell Infusion in Refractory/Relapsed Acute Myeloid Leukemia and Myelodysplastic Syndrome:The BigEMINy Study
Brief Title: Haploidentical Stem Cell Transplant With or Without NK Cell Infusion in AML and MDS
Acronym: Bigeminy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2588
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplasia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo-stem cell transplant followed by NK infusion (Experimental): Haplo stem cell transplant (from bone marrow or apheresis) is followed by a haplo-NK cell infusion (target dose ≥1*106/kg b.w.) at day 7.
  Unstimulated haplo-NK cells are collected through apheresis Mononuclear cells are then subjected to a preliminary negative selection of CD3+ cells and to a subsequent positive selection of CD56+ cells. CD3 negative/CD56 positive cells are infused
  Interventions: Biological: Haplo SCT with NK cells
- Haplo-stem cell transplant (Active Comparator): Patients in this arm receive standard haplo stem cell transplant (from bone marrow or apheresis) transplant without subsequent NK cell infusion.
  Interventions: Biological: Haplo SCT

INTERVENTIONS:
Biological: Haplo SCT with NK cells — Patients in this arm receive haplo-SCT followed by one boost of NK cells one/two weeks after the transplant. Lymphocyte are collected by apheresis from the donor one-two weeks after BM harvest. CD3 negative/CD56 positive cells are selected by immunomagnetic columns (other lymphocytes are stored to be used as DLI)
  Other Names: haplo SCT followed by NK cell infusion
  Arms: Haplo-stem cell transplant followed by NK infusion
Biological: Haplo SCT — Patients in this arm receive a standard haplo-SCT. All administerd therapies are the same as in other arm, except for the NK cell boost..
  Other Names: Standard haplo SCT without subsequent NK cell boost.
  Arms: Haplo-stem cell transplant

SUMMARY:
Relapse after an allogeneic hematopoietic stem cell transplantation (HSCT) is high in patients with advanced AML, in the 50% range. NK cells have been shown to possess significant anti-leukemic activity and may be used to reduce the incidence of relapse in patients with advanced AML.

Investigators hypothesize that the administration of a purified boost of NK cells on day +7 post HSCT, will reduce the incidence of relapse from the current 50% to 25%. In a phase III multicenter clinical study, 116 patients will be randomized to receive or not a boost of donor NK cells on day +7 post-HSCT. The first 10 patients in the experimental arm will be analyzed for toxicity. The stopping rule will be a transplant related mortality of more than 50% in the first 20 patients who received NK cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML or MDS
* Patients not in remission at the time of transplant
* Age 18-75
* ECOG performance status <2
* Availability of a family HLA haploidentical donor, eligible to donate both marrow cells and unstimulated lymphocytes (1 apheresis procedure at day +7) .

Exclusion Criteria:

* Positive serologic markers for human immunodeficiency virus (HIV)
* Acute hepatitis B virus (HBV) or acute hepatitis C virus (HCV) infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Leukemia relapse | 1 year after bone marrow transplant
  Cumulative incidence of leukemia relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bacigalupo, Prof, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy